CLINICAL TRIAL: NCT01218165
Title: The Inflammaging Network: Bridging Low Grade Inflammation With Gut Microbiota and Intestinal Barrier Function in Elderly Humans
Brief Title: Low Grade Inflammation, Gut Microbiota and Barrier Function in Elderly Humans
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Luzia Valentini, Research Scientist, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EA1/062/10
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Aged; Healthy
Keywords: Healthy Eldery People
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): without intervention
  Interventions: Other: Control Group
- Intervention Group (Experimental): This group receives a probiotic drink daily for 6 week.
  Interventions: Dietary Supplement: Probiotic drink

INTERVENTIONS:
Dietary Supplement: Probiotic drink — This group receives a probiotic drink daily for 6 week.
  Arms: Intervention Group
Other: Control Group — without intervention
  Arms: Control Group

SUMMARY:
Cardiovascular diseases (CVD) are the main cause of death in the European Union. A large part of the aging process, including immunosenescence, is explained by an imbalance between inflammatory and anti-inflammatory networks, wich results in the low grade chronic pro-inflammatory status termed inflammaging. It can contribute to a number of age-related chronic diseases (e.g. atherosclerosis, type 2 diabetes, Alzheimer disease, osteoporosis). Prevention or delay in onset of chronic diseases can potentially benefit a large segment of the elderly population. Now it is hypothesised that a probiotic drink can reduce low-grade inflammation through improvement of the gut barrier function and gut microbiota composition in elderly people with low-grade inflammation.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) are the main cause of death in the European Union. A large part of the aging process, including immunosenescence, is explained by an imbalance between inflammatory and anti-inflammatory networks, wich results in the low grade chronic pro-inflammatory status termed inflammaging. It can contribute to a number of age-related chronic diseases (e.g. atherosclerosis, type 2 diabetes, Alzheimer disease, osteoporosis). Prevention or delay in onset of chronic diseases can potentially benefit a large segment of the elderly population. Now it is hypothesised that a probiotic drink can reduce low-grade inflammation through improvement of the gut barrier function and gut microbiota composition in elderly people with low-grade inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Men >65 years of age.
* Body mass index: 22-34,9 kg/m²
* non-smokers

Intervention trial:

* hsCRP > 1 mg/L (Screening blood test)
* normal blood count (Screening blood test)
* normal ALAT, ASAT and serum creatinine levels (Screening blood test)

Exclusion Criteria:

* any major non-organic disease, including malign diseases (haematological, inflammatory, metabolic,)
* any major organ disease, including neoplastic diseases.
* intake of antibiotics within the last 6 weeks
* chronic therapy with analgetics (incl. acetylsalicylic acid)
* chronic therapy with proton pump inhibitors
* regular intake of probiotic bacteria products within the last 3 weeks
* chronic anti-inflammatory therapy with NSARs or previous therapy within the last 20 days
* subjects with expected non-compliance to protocol guidelines
* subjects that participate in other trials

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Pre/post-intervention change in hsCRP | 6 weeks
  Change (reduction) of hsCRP over a 6-week period in older persons.

SECONDARY OUTCOMES:
Intestinal permeability | 6 weeks
  Intestinal permeability tests will be performed with a triple sugar test (5 g LAC, 10 g MAN, and 20 g SAC dissolved in 100 ml of water).
Stool: Stool: Real-Time-PCR | 6 weeks
  During screening and post intervention quantitative Real-Time-PCR of bacterial 16S ribosomal RNA from feces will be performed.
Blood screening | 6 weeks
  Day 0 - Screening: hsCRP, leukocytes, erythrocytes, haemoglobin, haematokrit, sodium, potassium, glucose, total cholesterol, HDL, LDL, bilirubin total, bilirubin direct, ASAT, ALAT, creatinine Day 42 - post intervention: hsCRP, leukocytes, erythrocytes, haemoglobin, haematokrit, glucose, total cholesterol, HDL, LDL.
Muscle function | 6 weeks
  Handgrip strength will be evaluated using the Jamar vigorimeter (Preston, Jackson, MI 49204, USA) on Day 0 in the screening period and at the end of the intervention trial.
Physical performance status | 6 weeks
  The short physical performance battery (SPPB) (24) will be performed at the start and at the end of the intervention trial. SPPB is used to assess lower extremity function. It evaluates balance, gait, strength, and endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Luzia Valentini, Doctor, Principal Investigator — Charite University, Berlin, Germany; Herbert Lochs, Professor, Principal Investigator — Medical University of Innsbruck; Jörg-Dieter Schulzke, Professor, Principal Investigator — Charite University, Berlin, Germany; Stefan Bereswill, Professor, Principal Investigator — Charite University, Berlin, Germany; Alexander Swidsinski, Doctor, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Franceschi C, Capri M, Monti D, Giunta S, Olivieri F, Sevini F, Panourgia MP, Invidia L, Celani L, Scurti M, Cevenini E, Castellani GC, Salvioli S. Inflammaging and anti-inflammaging: a systemic perspective on aging and longevity emerged from studies in humans. Mech Ageing Dev. 2007 Jan;128(1):92-105. doi: 10.1016/j.mad.2006.11.016. Epub 2006 Nov 20. PMID 17116321
- [Background] Ballantyne CM, Nambi V. Markers of inflammation and their clinical significance. Atheroscler Suppl. 2005 May;6(2):21-9. doi: 10.1016/j.atherosclerosissup.2005.02.005. PMID 15823493
- [Background] Pearson TA, Mensah GA, Alexander RW, Anderson JL, Cannon RO 3rd, Criqui M, Fadl YY, Fortmann SP, Hong Y, Myers GL, Rifai N, Smith SC Jr, Taubert K, Tracy RP, Vinicor F; Centers for Disease Control and Prevention; American Heart Association. Markers of inflammation and cardiovascular disease: application to clinical and public health practice: A statement for healthcare professionals from the Centers for Disease Control and Prevention and the American Heart Association. Circulation. 2003 Jan 28;107(3):499-511. doi: 10.1161/01.cir.0000052939.59093.45. No abstract available. PMID 12551878
- [Background] Imhof A, Frohlich M, Loewel H, Helbecque N, Woodward M, Amouyel P, Lowe GD, Koenig W. Distributions of C-reactive protein measured by high-sensitivity assays in apparently healthy men and women from different populations in Europe. Clin Chem. 2003 Apr;49(4):669-72. doi: 10.1373/49.4.669. No abstract available. PMID 12651827
- [Background] Lannergard A, Friman G, Ewald U, Lind L, Larsson A. Serum amyloid A (SAA) protein and high-sensitivity C-reactive protein (hsCRP) in healthy newborn infants and healthy young through elderly adults. Acta Paediatr. 2005 Sep;94(9):1198-202. doi: 10.1111/j.1651-2227.2005.tb02074.x. PMID 16279005
- [Background] Libby P, Okamoto Y, Rocha VZ, Folco E. Inflammation in atherosclerosis: transition from theory to practice. Circ J. 2010 Feb;74(2):213-20. doi: 10.1253/circj.cj-09-0706. Epub 2010 Jan 9. PMID 20065609
- [Background] Pradhan AD, Manson JE, Rifai N, Buring JE, Ridker PM. C-reactive protein, interleukin 6, and risk of developing type 2 diabetes mellitus. JAMA. 2001 Jul 18;286(3):327-34. doi: 10.1001/jama.286.3.327. PMID 11466099
- [Background] Griffin WS. Inflammation and neurodegenerative diseases. Am J Clin Nutr. 2006 Feb;83(2):470S-474S. doi: 10.1093/ajcn/83.2.470S. PMID 16470015
- [Background] Kimble RB, Matayoshi AB, Vannice JL, Kung VT, Williams C, Pacifici R. Simultaneous block of interleukin-1 and tumor necrosis factor is required to completely prevent bone loss in the early postovariectomy period. Endocrinology. 1995 Jul;136(7):3054-61. doi: 10.1210/endo.136.7.7789332.
- [Background] Pirlich M, Norman K, Lochs H, Bauditz J. Role of intestinal function in cachexia. Curr Opin Clin Nutr Metab Care. 2006 Sep;9(5):603-6. doi: 10.1097/01.mco.0000241671.09676.d8. PMID 16912557
- [Background] D'Souza T, Sherman-Baust CA, Poosala S, Mullin JM, Morin PJ. Age-related changes of claudin expression in mouse liver, kidney, and pancreas. J Gerontol A Biol Sci Med Sci. 2009 Nov;64(11):1146-53. doi: 10.1093/gerona/glp118. Epub 2009 Aug 19. PMID 19692671
- [Background] Saltzman JR, Kowdley KV, Perrone G, Russell RM. Changes in small-intestine permeability with aging. J Am Geriatr Soc. 1995 Feb;43(2):160-4. doi: 10.1111/j.1532-5415.1995.tb06382.x. PMID 7836641
- [Background] Beaumont DM, Cobden I, Sheldon WL, Laker MF, James OF. Passive and active carbohydrate absorption by the ageing gut. Age Ageing. 1987 Sep;16(5):294-300. doi: 10.1093/ageing/16.5.294. PMID 3120502
- [Background] Guarner F. Enteric flora in health and disease. Digestion. 2006;73 Suppl 1:5-12. doi: 10.1159/000089775. Epub 2006 Feb 8. PMID 16498248
- [Background] Ordovas JM, Mooser V. Metagenomics: the role of the microbiome in cardiovascular diseases. Curr Opin Lipidol. 2006 Apr;17(2):157-61. doi: 10.1097/01.mol.0000217897.75068.ba. PMID 16531752
- [Background] Turnbaugh PJ, Ridaura VK, Faith JJ, Rey FE, Knight R, Gordon JI. The effect of diet on the human gut microbiome: a metagenomic analysis in humanized gnotobiotic mice. Sci Transl Med. 2009 Nov 11;1(6):6ra14. doi: 10.1126/scitranslmed.3000322. PMID 20368178
- [Background] Degens H. Age-related skeletal muscle dysfunction: causes and mechanisms. J Musculoskelet Neuronal Interact. 2007 Jul-Sep;7(3):246-52. PMID 17947808
- [Background] Hamer M, Molloy GJ. Association of C-reactive protein and muscle strength in the English Longitudinal Study of Ageing. Age (Dordr). 2009 Sep;31(3):171-7. doi: 10.1007/s11357-009-9097-0. Epub 2009 May 23. PMID 19466582
- [Background] Schaap LA, Pluijm SM, Deeg DJ, Visser M. Inflammatory markers and loss of muscle mass (sarcopenia) and strength. Am J Med. 2006 Jun;119(6):526.e9-17. doi: 10.1016/j.amjmed.2005.10.049. PMID 16750969
- [Background] Goebel A, Buhner S, Schedel R, Lochs H, Sprotte G. Altered intestinal permeability in patients with primary fibromyalgia and in patients with complex regional pain syndrome. Rheumatology (Oxford). 2008 Aug;47(8):1223-7. doi: 10.1093/rheumatology/ken140. Epub 2008 Jun 7. PMID 18540025
- [Background] Swidsinski A, Loening-Baucke V, Verstraelen H, Osowska S, Doerffel Y. Biostructure of fecal microbiota in healthy subjects and patients with chronic idiopathic diarrhea. Gastroenterology. 2008 Aug;135(2):568-79. doi: 10.1053/j.gastro.2008.04.017. Epub 2008 Apr 18. PMID 18570896
- [Background] Swidsinski A, Weber J, Loening-Baucke V, Hale LP, Lochs H. Spatial organization and composition of the mucosal flora in patients with inflammatory bowel disease. J Clin Microbiol. 2005 Jul;43(7):3380-9. doi: 10.1128/JCM.43.7.3380-3389.2005. PMID 16000463
- [Background] Swidsinski A. Standards for bacterial identification by fluorescence In situ hybridization within eukaryotic tissue using ribosomal rRNA-based probes. Inflamm Bowel Dis. 2006 Aug;12(8):824-6; author reply 826-7. doi: 10.1097/00054725-200608000-00018. No abstract available. PMID 16917237
- [Background] Puthoff ML, Janz KF, Nielson D. The relationship between lower extremity strength and power to everday walking behaviors in older adults with functional limitations. J Geriatr Phys Ther. 2008;31(1):24-31. doi: 10.1519/00139143-200831010-00005. PMID 18489805